CLINICAL TRIAL: NCT03811899
Title: 18F-DCFPyL PET/CT in High-grade Epithelial Ovarian Cancer
Brief Title: 18F-DCFPyL PET/CT in High-grade Epithelial Ovarian Cancer (PET HOC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-6241
Record Dates: First submitted 2019-01-08; First posted 2019-01-22 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Stage III Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm study to determine whether HG EOC are 18F-DCFPyL-avid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL PET/CT imaging (Experimental): We will use technology called PET-CT that combines a Positron Emission Tomography (PET) scan with a computed tomography (CT) scan. This combined imaging test, where PET and CT data is gathered at one time, will be performed on an integrated PET-CT scanner located at Princess Margaret Cancer Centre.
  Interventions: Diagnostic Test: 18F-DCFPyL

INTERVENTIONS:
Diagnostic Test: 18F-DCFPyL — The purpose of this study is to determine whether HG SOC are 18F-DCFPyL (=GCP-II)-avid and to compare the performance of this PET to CT and findings at time of surgery.

SUMMARY:
The purpose of this study is to determine whether high grade epithelial ovarian cancers (=HG EOC) are 18F-DCFPyL (=2-(3-(1-carboxy-5-[(6-[18F]fluoro-pyridine-3-carbonyl)-amino]-pentyl)-ureido)-pentanedioic acid)-avid and to compare the performance of this PET to CT and findings at time of surgery

Background:

There is a need for better noninvasive tools that will map disease extent in HG EOC. A recent study has shown that at immunohistochemistry GCP=II is overexpressed in ovarian cancer tumors, both primary and metastatic. Glucose carboxypeptidase-II (=GCP-II), also known as prostate specific membrane antigen (= PSMA) has been used clinically to assess patients with prostate cancer and many other tumors have been shown to be PSMA-avid on PET (including renal cell carcinomas).

18F-DCFPyL has the potential to improve patient selection for primary therapy. If successful, this may decrease the rate of futile surgeries and associated morbidity and better direct patients to the most appropriate therapy primary debulking surgery (PDS) vs neoadjuvant chemotherapy (NACT). Furthermore, if high-level GCP-II expression is shown at preoperative imaging in patients with HG EOC, this may be used in considering feasibility of future theranostic applications.

Study Design:

This is a single arm pilot study to assess whether HG EOC are 18F-DCFPyL-avid.

In this prospective trial, the investigators will recruit 20 women whom will undergo conventional staging with contrast-enhanced CT of the abdomen and pelvis as per standard of care. All disease sites, primary and metastatic will be recorded using a standardized reporting template.

Subsequently, 18F-DCFPyL-PET/CT will be performed (within 6 weeks of CT).

All disease sites on PET will be recorded using same reporting template in addition to qualitative and semiquantitative evaluation (SUV measurement) of all known tumor sites.

DETAILED DESCRIPTION:
In patients with ovarian cancer, identifying the volume and exact locations of disease is of paramount importance prior to deciding on upfront surgery versus chemotherapy. Currently, most clinicians use CT scans to determine the extent of disease; however, this tool has limited sensitivity and specificity. 18F-Fluorodeoxyglucose (=FDG) PET scans have been previously assessed with only limited success; therefore, FDG PET scans have not been universally incorporated into the workup of patients with ovarian cancer. A further noninvasive tool that would accurately map disease extent is needed to better select therapy for ovarian cancer patients, reduce the rate of aborted surgery and associated complications, and hopefully improve overall outcome.

"Glutamate carboxypeptidase II (GCP-II)" is a type of an enzyme on the surface of cells. It has additional names including prostate specific membrane antigen (PSMA). It is expressed by normal tissues such as salivary glands, as well as by multiple malignant tumors, often in the abnormal blood vessels of these tumors. A recent study has examined the expression of this enzyme in gynecologic cancers including primary and metastatic ovarian cancer. The authors showed a high expression of this enzyme at special staining performed on surgical tumor samples. In other cancers, such as prostate cancer PET with GCP-II (=PSMA PET) has shown very high sensitivity and high specificity for the detection of tumor sites, even when CT is negative. In this study the investigators will be assessing the performance of this special PET scan using a PSMA tracer called "18F-DCFPyL". The investigators will investigate the ability of 18F-DCFPyL PET scans to detect sites of disease in patients with ovarian cancer. Disease sites seen on PET will be compared to what is seen on the standard CT scan, and to what is found at time of surgery (if surgery is performed).

The rationale for this study is that there is a need for better noninvasive tools that will map disease extent in HG EOC. A recent study has shown that at immunohistochemistry GCP=II is overexpressed in ovarian cancer tumors, both primary and metastatic. GCP-II (=PSMA) has been used clinically to assess patients with prostate cancer and many other tumours have been shown to be PSMA-avid on PET (including renal cell carcinomas). The purpose of this study is to determine whether HG SOC are 18F-DCFPyL (=GCP-II)-avid and to compare the performance of this PET to CT and findings at time of surgery.

Primary Objective

To determine whether HG EOCs are 18F-DCFPyL avid on PET/CT.

Secondary Objectives:

To compare the sites of disease identified on PET/CT to contrast-enhanced CT (standard of care).

To determine whether there is heterogeneity in 18F-DCFPyL-avidity at different tumor sites.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Cytological or histological diagnosis of high grade epithelial ovarian cancer, or clinical suspicious of HG EOC based on symptoms, physical exam, tumor markers and imaging findings.
* Clinical stage III or IV, being considered for primary debulking surgery or NACT.
* Contrast-enhanced CT abdomen and pelvis within 6 weeks of PET (prior to enrollment).

Exclusion Criteria:

* Inability to provide informed consent.
* Contraindication for PET examination as per institutional safety guidelines, including but not limited to pregnancy, or inability to lie still for PET examination.
* Evidence of the following epithelial ovarian cancer histological subtypes: Mucinous, low grade serous, low grade endometrioid and low-malignant potential tumors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
18F-DCFPyL-avid PET/CT | Through study completion up to 2 years
  To determine the proportion of HG EOC that are18F-DCFPyL-avid on PET/CT.

SECONDARY OUTCOMES:
18F-DCFPyL PET/CT vs. Contrast-enhanced CT | Through study completion up to 2 years
  The determine the proportion of HG EOC tumor sites detected on 18F-DCFPyL PET/CT compared to contrast-enhanced CT

CONTACTS AND LOCATIONS:
Overall Officials: Ur Metser, MD, Principal Investigator — UHN
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kunikowska J, Bizon M, Pelka K, Derlatka P, Olszewski M, Krolicki L. 68 Ga-Prostate-Specific Membrane Antigen PET/CT in Ovarian Tumors : Potential to Differentiate Benign and Malignant Tumors Before Surgery: A Preliminary Report. Clin Nucl Med. 2023 Feb 1;48(2):e60-e66. doi: 10.1097/RLU.0000000000004486. Epub 2022 Nov 18. PMID 36512649
- [Derived] Metser U, Kulanthaivelu R, Chawla T, Johnson S, Avery L, Hussey D, Veit-Haibach P, Bernardini M, Hogen L. 18F-DCFPyL PET/CT in advanced high-grade epithelial ovarian cancer: A prospective pilot study. Front Oncol. 2022 Oct 13;12:1025475. doi: 10.3389/fonc.2022.1025475. eCollection 2022. PMID 36313720